CLINICAL TRIAL: NCT04548362
Title: Biomarkers of Meats and Potatoes Intake: a Meal Study in Healthy Men and Women - the MEPO Study
Brief Title: Biomarkers of Meats and Potatoes Intake
Acronym: MEPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Professor Lars Ove Dragsted (Other)
Responsible Party: Sponsor-Investigator, Professor Lars Ove Dragsted, Professor, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: H-150204011H
Record Dates: First submitted 2020-09-07; First posted 2020-09-14 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Nutrition Disorders
Keywords: Biomarkers of food intake
MeSH Terms: conditions — Nutrition Disorders

STUDY DESIGN:
Intervention Model Description: Subjects were randomised to four meals with meats and starchy foods in such a way that all volunteers had each meat and each starchy food once and so that all combinations of meats and starchy foods were equally common. Each volunteer was also randomised to the sequence of the meals.
Masking Description: It is not possible to mask foods and for the explorative analysis of results, masking is not required.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meat meals (Experimental): This arm contains a 4-way cross-over intervention study with meats
  Interventions: Other: Meat arm
- Starchy meals (Experimental): This arm contains a 4-way cross-over intervention study with
  Interventions: Other: Starchy foods arm

INTERVENTIONS:
Other: Meat arm — Randomised sequence of pork, beef, chicken meat, and an egg white/pea combination
  Arms: Meat meals
Other: Starchy foods arm — Randomised sequence of boiled potato, fried potato, potato crisps, and boiled white rice
  Arms: Starchy meals

SUMMARY:
This cross-over meal study is a four-way intervention with 12 volunteers randomized at the same time to four meals with fried meats (beef, pork, chicken and amino-acid matched non-meat control) and to four meals with potato products (boiled, chips, fries, and a control with boiled white rice) to search for biomarkers of intake.

DETAILED DESCRIPTION:
In a two-dimensional, cross-over meal study, 12 healthy volunteers consumed in a randomized sequence four test meals: chicken, pork, beef, and a control made of egg white and pea. At the same time they were independently randomized to four starchy foods to be consumed together with the meats: boiled potatoes, fried potatoes, potato crisps or boiled white rice. Fasting and postprandial urine samples were collected to cover 48 h after each meal and samples were profiled by untargeted LC-ESI-qTOF-MS metabolomics. The profiles following the meal challenges were explored by univariate and multivariate analyses and single and combined markers of intake identified chemically by MS/MS fragmentation experiments and statistically by ROC curves and error rates as well as FDR statistics.

ELIGIBILITY:
Inclusion Criteria:

* healthy

Exclusion Criteria:

* non-pregnant, no abuse of alcohol or drugs, no chronic medication except p-pills

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-02-15 (Actual); Primary Completion 2016-05-30 (Actual); Study Completion 2016-05-30 (Actual)

PRIMARY OUTCOMES:
meat intake biomarkers | 0-48 hours
  To identify intake biomarkers of general meat, red meat and poultry
Potato intake biomarkers | 0-48 hours
  To identify intake biomarkers of general potato, fried potato and white rice

CONTACTS AND LOCATIONS:
Overall Officials: Catalina Cuparencu, PhD, Study Director — University of Copenhagen
Locations (1):
- Lars Dragsted, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Adding samples to CUBE (www.cube.ku.dk), supporting information to the ERDA sharing system, and sample database and study data to the DASH-IN database for data sharing.
Supporting Information: Study Protocol, ICF
Time Frame: 1 year
Access Criteria: after contact with PI; only anonymized information will be provided.

REFERENCES:
- [Background] Zhou X, Ulaszewska MM, Cuparencu C, De Gobba C, Vazquez-Manjarrez N, Gurdeniz G, Chen J, Mattivi F, Dragsted LO. Urine Metabolome Profiling Reveals Imprints of Food Heating Processes after Dietary Intervention with Differently Cooked Potatoes. J Agric Food Chem. 2020 Jun 3;68(22):6122-6131. doi: 10.1021/acs.jafc.0c01136. Epub 2020 May 8. PMID 32338001
- [Result] Cuparencu C, Rinnan A, Dragsted LO. Combined Markers to Assess Meat Intake-Human Metabolomic Studies of Discovery and Validation. Mol Nutr Food Res. 2019 Sep;63(17):e1900106. doi: 10.1002/mnfr.201900106. Epub 2019 Jun 13. PMID 31141834